CLINICAL TRIAL: NCT03814759
Title: Preoperative S-1 Plus Cisplatin-based Chemoradiotherapy for Locally Advanced Resectable Gastric Adenocarcinoma : Randomized, Phase II Trial
Brief Title: Preoperative Chemoradiotherapy for Locally Advanced Resectable Gastric Adenocarcinoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Principal Investigator, Hyo Song Kim, professor, Yonsei University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 4-2015-0603
Record Dates: First submitted 2019-01-23; First posted 2019-01-24 (Actual); Last update posted 2024-12-27 (Actual); Status verified 2021-04

CONDITIONS: Gastric Adenocarcinoma
MeSH Terms: interventions — titanium silicide; Cisplatin; Radiation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- SP+CCRT (Experimental): S-1 20mg/m2, bid (D1~14, D22~35) Cisplatin 30mg/m2/day (W1, 2, 4, 5) radiation 45Gy per 5 weeks
  Interventions: Drug: TS-1 + cisplatin; Radiation: radiation

INTERVENTIONS:
Drug: TS-1 + cisplatin — S-1 20mg/m2, bid (D1~14, D22~35) Cisplatin 30mg/m2/day (W1, 2, 4, 5)
Radiation: radiation — radiation 45Gy per 5 weeks

SUMMARY:
Gastric cancer is a high incidence in Asia, and one of the leading cause of death in Korea. A cure rate is improving due to early diagnosis. However, the 5-year survival rate of gastric cancer excluding early gastric cancer is about 40 ~ 67%. Therefore, several methods for lowering the recurrence rate have been attempted and concurrent chemoradiotherapy can be considered as a method to lower the recurrence rate of gastric cancer. The purpose of this study is to evaluate the pathologic response rate and safety of patients who underwent surgery after chemoradiotherapy.

DETAILED DESCRIPTION:
Gastric cancer is a high incidence in Asia, and one of the leading cause of death in Korea. A cure rate is improving due to early diagnosis. However, the 5-year survival rate of gastric cancer excluding early gastric cancer is about 40 ~ 67%. Therefore, several methods for lowering the recurrence rate have been attempted and concurrent chemoradiotherapy can be considered as a method to lower the recurrence rate of gastric cancer. The purpose of this study is to evaluate the pathologic response rate and safety of patients who underwent surgery after chemoradiotherapy.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 20 years old
2. Histologically confirmed gastric adenocarcinoma
3. clinical stage : resectable gastric cancer

   * advanced confirmed (EGD)
   * extramural infiltration> 1 mm (CT)
   * positive serosa invasion (EUS)
4. Eastern Cooperative Oncology Group performance status 0 or 1
5. no prior chemotherapy and radiotherapy
6. measurable lesion or evaluable lesion according to Response Evaluation Criteria in Solid Tumors version 1.1 criteria
7. Patients with adequate organ function
8. Signed informed consent

Exclusion Criteria:

1. Metastasis esophageal invasion > 3cm
2. inoperable peritoneal seeding disease determined by exploratory laparotomy
3. T4b invading the surrounding organs
4. lymph node metastasis outside the celiac trunk Lymph node and splenic lymph node
5. uncontrolled viral infections (HIV, HBV, HCV)
6. Pregnant or lactating women, women of childbearing potential not employing adequate contraception
7. severe hypersensitivity reactions to S-1, cisplatin
8. Subjects with uncontrolled clinically significant cardiovascular medical history, uncontrolled infection or complication
9. Other co-existing malignancies or malignancies diagnosed within the last 5 years except for curatively treated non-melanoma skin cancer or in situ carcinoma of the cervix

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2016-12-12 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2022-07-31 (Actual)

PRIMARY OUTCOMES:
pathological response rate | 10 week
  to evaluate pathological response rate in locally advanced resectable gastric cancer

CONTACTS AND LOCATIONS:
Locations (1):
- Severance Hospital, Yonsei University Health System, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No